CLINICAL TRIAL: NCT06627244
Title: Phase 2, Single Arm Study of Tebentafusp and Radioembolization in the Treatment of Metastatic Uveal Melanoma
Brief Title: Study of Tebentafusp and Radioembolization in the Treatment of Metastatic Uveal Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Immunocore Ltd (Industry)
Responsible Party: Principal Investigator, Lynn Feun, MD, Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20231324
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Uveal Melanoma; Metastatic Uveal Melanoma in the Liver
MeSH Terms: conditions — Uveal Melanoma | interventions — tebentafusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Tebentafusp in combination with Radioembolization Group (Experimental): Participants in this group will first be administered Yttrium 90 Trans-Arterial Radioembolization (Y90 TARE) therapy, followed by a 14 to 28 day recovery period. Participants will then be administered Tebentafusp once weekly during every 28-day cycle. Participants may receive up to 24 months or 24 cycles of Tebentafusp therapy.
  Total participation is about 3 years.
  Interventions: Drug: Tebentafusp; Radiation: TheraSphere™ Yttrium-90 Trans-Arterial Radioembolization

INTERVENTIONS:
Drug: Tebentafusp — Tebentafusp will be administered intravenously to participants at or within 28 days of their first Y-90 TARE procedure. This 28-day period includes the 14- to 28-day Y-90 TARE Recovery Period. For administrative purposes, one cycle of tebentafusp treatment is 28 days in length. Tebentafusp will be administered on a dose escalation schedule for Cycle 1 starting at 20 mcg on Day 1, increasing to 30 mcg on Day 8, and a final dose of 68 mcg on Day 15, which will be administered once per week until unacceptable toxicity develops, disease progression, or withdrawal of consent, whichever occurs first.
  Other Names: Tebentafusp-tebn
Radiation: TheraSphere™ Yttrium-90 Trans-Arterial Radioembolization — Participants will undergo radiographic and 99mTC-labeled macroaggregated albumin (99mTc-MAA) assessment for suitability prior to Y-90 absorbed glass microsphere treatment per institutional procedures. Y-90 trans-arterial radioembolization (TARE) is a standard of care treatment for intrahepatic metastases of uveal melanoma as indicated in the National Comprehensive Cancer Network (NCCN) consensus guidelines (NCCN Guidelines®, 2023). Y-90 absorbed glass microspheres will be administered at least one time prior to initiating Tebentafusp treatment. After the Y90-TARE procedure, participants will have a 14- to 28-day Y-90 TARE Recovery Period.
  Other Names: Y-90 TARE

SUMMARY:
The purpose of this study is to determine the effects (good and bad) that Tebentafusp in combination with Yttrium-90 (Y-90) radioembolization has on patients with metastatic uveal melanoma that has spread to the liver.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic uveal melanoma, confined mainly to the liver, and documented by pathology review
2. Serum bilirubin <2 mg/dl, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 5 x upper limit of normal (ULN)
3. Mapping angiogram procedure shows radioembolization is feasible and safe to perform
4. Human leukocyte antigen-A*02:01(HLA A⁕ 02:01) positive
5. Patient age ≥ 18 years old
6. Ability to provide and understand written informed consent
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
8. Patients must have measurable disease or non-measurable disease according to RECIST 1.1 (Eisenhauer et al, 2009).

Exclusion Criteria:

1. Patient with any tumor size > 8 cm
2. Total bilirubin > 1.5 × ULN, except for patients with Gilbert's syndrome, who are excluded if total bilirubin > 3.0 × ULN or direct bilirubin > 1.5 × ULN
3. Clinical laboratory measurements that meet any of the following criteria:

   * Alanine aminotransferase (ALT) > 3 × ULN
   * Aspartate aminotransferase (AST) > 3 × ULN
   * Absolute neutrophil count (ANC) < 1.0 × 10^9 cells/L
   * Absolute lymphocyte count < 0.5 × 10^9 cells/L
   * Platelet count < 75 × 109 platelets/L
   * Hemoglobin < 8 g/dL
4. Angiogram shows vascular shunting which prevents radioembolization
5. History of severe hypersensitivity reactions (eg, anaphylaxis) to other biologic drugs or monoclonal antibodies
6. Patients with clinically significant cardiac disease or impaired cardiac function, including any of the following:

   * Congestive heart failure (New York Heart Association Class ≥ 3).
   * Uncontrolled hypertension (consistent findings of systolic blood pressure [BP] > 160 mmHg or diastolic BP > 110 mmHg).
   * History of ventricular arrhythmia currently requiring medical treatment.
   * Uncontrolled atrial fibrillation.
   * Electrocardiogram (ECG) QT interval corrected for heart rate by Fridericia's method (QTcF) > 470 msec during screening obtained on triplicate ECGs or known history of congenital prolonged QT syndrome.
   * Acute myocardial infarction or unstable angina pectoris ≤ 6 months prior to screening.
7. Presence of symptomatic or untreated central nervous system (CNS) metastases or CNS metastases that require doses of corticosteroids within 14 days prior to study treatment Day 1.
8. Active infection requiring systemic antibiotic therapy. Patients requiring systemic antibiotics for infection must have completed therapy at least 1 week prior to the first dose of Tebentafusp.
9. Known history of human immunodeficiency virus (HIV) infection. Testing for HIV status is not necessary unless clinically indicated.
10. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection per institutional protocol. Testing for HBV or HCV status is not necessary unless clinically indicated or the patient has a history of HBV or HCV infection.
11. Malignant disease other than that being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to study treatment; completely resected basal cell and squamous cell skin cancers; any malignancy considered to be indolent and that has never required therapy; and completely resected carcinoma in situ of any type.
12. Any medical condition that would, in the Investigator's or Sponsor's judgment, prevent the patient's participation in the clinical study due to safety concerns, compliance with clinical study procedures, or interpretation of study results
13. Patients who received systemic treatment with steroids or any other immunosuppressive drug within 2 weeks of the planned first dose of study intervention. The following exceptions are permitted (Section 4.9.1):

    * Treatment for well-controlled and asymptomatic adrenal insufficiency, but replacement dosing is limited to prednisone ≤ 12 mg daily or the equivalent.
    * Local steroid therapies (eg, optic, ophthalmic, intra-articular, or inhaled medications).
    * Premedication for allergy to contrast reagent.
    * Steroids for management of CNS metastases > 14 days prior to the planned first dose of study intervention.
    * To treat asthma or chronic obstructive pulmonary disease exacerbations > 14 days prior to the planned first dose of study intervention (only short-term oral or IV use in doses > 12 mg/day prednisone equivalent).
    * For inhalation in the management of asthma or chronic obstructive pulmonary disease.
    * Any premedications required per protocol.
14. Patient with morning cortisol < lower limit of normal (unless the participant has asymptomatic adrenal insufficiency and is receiving stable replacement doses). For additional information regarding patients with adrenal insufficiency.
15. History of interstitial lung disease
16. History of pneumonitis that required corticosteroid treatment or current pneumonitis
17. Patients with active autoimmune disease requiring immunosuppressive treatment, including inflammatory bowel disease (ulcerative colitis or Crohn's disease), within 2 years of screening. Note: The following exceptions are permitted:

    * Vitiligo
    * Alopecia
    * Managed hypothyroidism (on stable replacement doses)
    * Asymptomatic adrenal insufficiency (on stable replacement doses) (For additional information regarding patients with adrenal insufficiency.
    * Psoriasis
    * Resolved childhood asthma/atopy
    * Well-controlled asthma
    * Type I diabetes mellitus
18. Major surgery within 2 weeks of the first dose of study drug (minimally invasive procedures such as bronchoscopy, tumor biopsy, insertion of a central venous access device, and insertion of a feeding tube are not considered major surgery and are not exclusionary)
19. Radiotherapy within 2 weeks of the first dose of study drug, with the exception of palliative radiotherapy to a limited field, such as for the treatment of bone pain or a focally painful tumor mass
20. Use of hematopoietic colony-stimulating growth factors (eg, granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), macrophage colony-stimulating factor (M-CSF)) ≤ 3 weeks prior to start of Tebentafusp. An erythroid-stimulating agent is allowed as long as it was initiated at least 3 weeks prior to the first dose of study treatment and the patient is not red blood cell (RBC) transfusion dependent. For more information on the timing and use of hematopoietic colony-stimulating growth factors during study.
21. Patient receiving a live or attenuated vaccine(s) ≤ 28 days prior to the first dose of study intervention. Note: Non-live vaccines (including adenoviral and messenger ribonucleic acid (mRNA)-based coronavirus disease-2019 (COVID-19) vaccines) are allowed but are not to be administered for at least 2 weeks before and 3 weeks after start of study treatment and within 24 hours before or after study treatment administration following the first 3 weeks of study treatment.
22. Pregnant, likely to become pregnant, or lactating women (where pregnancy is defined as the state of a female after conception and until the termination of gestation)
23. Women of childbearing potential (WoCBP) who are sexually active with a non-sterilized male partner, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective contraception during study treatment (defined in Section 4.12), and must agree to continue using such precautions for 6 months after the final dose of Tebentafusp; cessation of birth control after this point should be discussed with a responsible physician. Highly effective methods of contraception are described in Section 4.12.
24. Male patients must be surgically sterile or use double barrier contraception methods as described in Section 4.12 from enrollment through treatment and for 6 months following administration of the last dose of Tebentafusp.
25. Prior radioembolization or other regional, liver-directed therapy, including chemotherapy or embolization to same site in the liver
26. Patients with impaired decision-making capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2028-02-17 (Estimated); Study Completion 2031-02-17 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 24 months
  Progression-free survival (PFS) will be defined as the elapsed time in months from the first date of study treatment until documented disease progression, per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or death from any cause, whichever is earlier. For participants who remain alive without progression, follow-up time will be censored at the date of last disease assessment.
Number of Participants Experiencing Treatment-Related Adverse Events | Up to 24 months
  The number of participants experiencing treatment-related adverse events (AEs) and serious adverse events (SAEs) in participants receiving protocol therapy will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5, per physician discretion.

SECONDARY OUTCOMES:
Disease control rate (DCR) measured by proportion of patients | Up to 24 months
  Disease control rate (DCR) is the proportion of patients whose best response per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria is complete response (CR), partial response (PR), or stable disease (SD) confirmed with new assessments by CT or MRI imaging prior to starting new anticancer therapies. Response recorded after non-protocol anticancer therapy will not be counted.
Overall response rate (ORR) | Up to 2 years
  Overall response rate (ORR) is the proportion of patients whose best overall response per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria is complete response (CR) or partial response (PR). Response recorded after non-protocol anticancer therapy will not be counted.
Duration of response (DOR) | Up to 24 months
  The duration of overall response (DOR) is measured from the time in months measurement criteria are met for complete response (CR) or partial response (PR) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). For participants without progression, follow-up time will be censored at the date of last disease assessment (as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1).
Overall survival (OS) | Up to 3 years
  Overall survival (OS) is defined as the elapsed time in years from date of first study treatment until death from any cause. Participants without documented death will be censored at the last date known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Feun, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No